CLINICAL TRIAL: NCT06581679
Title: Treatment of Infertile Adenomyosis Patients Using Levonorgestrel-releasing Intrauterine System or Gonadotropin-releasing Hormone Agonist Before Frozen Blastocyst Transfer Improves Manifestations and Increases the Chances of Pregnancy
Brief Title: Adenomyosis and Pregnancy: Levonorgestrel vs. GnRH for Blastocyst Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Elnagar, Assistant professor of Obstetrics & Gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB#506 11/8-2024
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The levonorgestrel-releasing intrauterine system Group (Active Comparator)
  Interventions: Device: levonorgestrel-releasing intrauterine system; Procedure: frozen embryo transfer
- GnRHa Group (Active Comparator)
  Interventions: Drug: Triptorelin; Procedure: frozen embryo transfer

INTERVENTIONS:
Drug: Triptorelin — GnRHa will be given as a subcutaneous injection of triptorelin in a dose of 3.75 mg monthly for three months.
  Arms: GnRHa Group
Device: levonorgestrel-releasing intrauterine system — The levonorgestrel-releasing intrauterine system releasing 20 levonorgestrel daily.
  Arms: The levonorgestrel-releasing intrauterine system Group
Procedure: frozen embryo transfer — Frozen embryo transfer (FET) where a previously frozen embryo is thawed and transferred into a woman's uterus.
  The FET process involves hormone preparation to prepare the uterus for the transfer, embryo thawing, and the actual transfer of the embryo into the uterus. If the embryo implants and develops successfully, pregnancy can occur.

SUMMARY:
Adenomyosis is a condition where endometrial tissue grows into the uterine muscle, causing symptoms like pelvic pain, heavy bleeding, and infertility. This abnormal growth can lead to a variety of reproductive issues, including a higher risk of miscarriage and early pregnancy loss.

While there are treatments available for adenomyosis, they are often limited due to the lack of precise diagnostic criteria. One common approach is the use of gonadotropin-releasing hormone agonist (GnRHa), which can improve pregnancy rates in infertile women with adenomyosis. However, it's important to note that GnRHa may not restore pregnancy rates to baseline levels.

Another potential treatment option is the levonorgestrel-releasing intrauterine system (LNG-IUS). This device releases a hormone called levonorgestrel into the uterus, which can help control the symptoms of endometriosis and adenomyosis. Studies have shown that the endometrial concentration of levonorgestrel from the LNG-IUS is significantly higher than in other tissues like the myometrium, fallopian tubes, and fat tissue.

ELIGIBILITY:
Inclusion Criteria:

* Women who have adenomyosis diagnostic characteristics and underwent ICSI that resulted in good-quality FE.

Exclusion Criteria:

* Women Women who have adenomyosis diagnostic characteristics and underwent ICSI that resulted in Poor-quality FE.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Adenomyosis Treatment | 6 monthes
  Proportion of patients reporting at least a 50% reduction in pain (measured by pain, Enjoyment, and General Activities score) post-Adenomyosis Treatment.
Increase in Chemical and Clinical Pregnancy Rates | 6 Months
  Proportion of patients reported with pregnancy after Frozen Embryo transfer which is assessed by finding Heartbeats in the Trans-vaginal Ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Ash Sharqia Governorate, Egypt